**Study Title:** Social Networks and Methadone Maintenance Treatment Retention and Antiretroviral Therapy Retention in Tanzania

**Document:** Statistical Analysis Plan (ID: IRB00019420)

NCT number: NCT04479475

**Document date:** 8/11/2025

PI Name: Haneefa Saleem

Study Title: Adaptation and Pilot of a Social Network Intervention to Improve Retention in

Medication-Assisted Treatment for Opioid Use Disorder in Tanzania

## **Data Analysis Plan**

## I. Descriptive Analyses

- a. Baseline characteristics
  - i. Summarize participant demographics (age, gender, education, housing status, employment status, etc.)
  - ii. Describe baseline clinical characteristics (confirmed HIV status, methadone dosage, missed methadone doses in the past 30 days, ART refills in the past 6 months (for participants with confirmed HIV-positive status)
  - iii. Statistics: Means (SD) and medians (IQR) for continuous variables, counts and percentages for categorical variables

## II. Primary outcomes: Acceptability and Feasibility

- i. Intervention completion rates and individual session attendance for enrolled MMT clients and social support persons. Number of participants lost to follow-up or number who voluntarily withdrew from the study.
- ii. Content or thematic analysis of implementation facilitators and barriers/challenges, including any protocol deviations, as reported in follow-up, qualitative interviews with participants and intervention counselors, as well as in supervision meetings throughout the intervention implementation period.
- iii. Reported fidelity from intervention counselors, as reported in supervision meetings throughout the intervention implementation period, as well as in follow-up, qualitative interviews with counselors.

## III. Secondary outcomes: Missed Methadone Doses and ART refills

- a. Secondary outcomes will be assessed for MMT client participants only.
- b. Change in missed methadone doses in the past 30 days: Use the Wilcoxon signed-rank test to compare the number of missed methadone doses at baseline and follow-up. Report the median differences, mean differences for changes in missed doses, and the exact p-value.
- c. Change in pharmacy ART refills in the past 6 months (HIV-positive participants only): Conduct cross-tabulation to compare ART refill status at baseline and follow-up. Use McNemar's test to examine changes in refill status across the two time points. Report the proportions of participants refilling ART, the odds ratio, and the exact p-value.